CLINICAL TRIAL: NCT00493350
Title: International Stage IV Stratification Study (ISSS): Prospective Validation Trial of Circulating Tumor Cells (CTCs) as Prognostic and Predictive Markers in Women With Metastatic Breast Cancer About to Start First-Line Treatment
Brief Title: Prospective Validation Trial of Circulating Tumor Cells (CTCs) in Women With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 2005-0278
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Circulating Tumor Cells; Gene Profiling; International Stage Stratification Study; Blood Sample; ISSS
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collected prior to the initiation of chemotherapy as follows: 1 x 4 ml (serum tube), 2x10 ml (CellSave Tube), and 1x10 ml EDTA (selected centers); To perform global gene profiling on selected specimens and correlate the profiles with clinical outcomes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with newly diagnosed stage IV breast cancer scheduled to start systemic therapy.
  Interventions: Procedure: Blood Sample

INTERVENTIONS:
Procedure: Blood Sample — 1x4 ml (Serum Tube); 2x10 ml (CellSave Tube); 1x10 ml EDTA (Selected Centers)

SUMMARY:
Primary Objectives:

1. To validate the prognostic significance of circulating tumor cells (CTCs) in patients with newly diagnosed metastatic breast cancer (MBC).
2. To prospectively determine if assessment of CTCs can be used to stratify patients with MBC into two prognostic groups independent of existing methods i.e. hormone-receptor status, site of metastasis (e.g. visceral vs. non visceral) and treatment administered (e.g. chemotherapy vs. hormonal therapy).
3. To incorporate this information into the current TNM staging system by sub-classifying stage IV disease into two prognostic groups, Stage IVA and Stage IVB.

Secondary Objective:

1. To perform global gene profiling on selected specimens and correlate the profiles with clinical outcomes.

DETAILED DESCRIPTION:
Patients with tumors that have spread to other parts of the body and who are about to start systemic treatment will be eligible to take part in this study.

As is standard of care, you will have an evaluation of your disease through CT scans, bone scans, and PET scans. Before you begin your routine treatment, participants in this study will have 3 teaspoons of blood drawn at an M. D. Anderson clinic. This will be the only blood draw required for this study. You will then begin receiving standard therapy for your disease as decided by your treating physician.

You will have follow-ups with either your physician or through the research personnel (by phone calls by the research nurse) at 3, 6, 12, 18, and 36 months. After 36 months, follow-up will continue indefinitely at your doctor's discretion. At these follow-ups, your medical record will be reviewed to gather information for this study.

One of the blood samples will be preserved and used for research and development purposes specifically related to this study. This research includes also analysis of the tumor gene profiling. This study will be done to better understand the biology of metastatic breast cancer. Neither participants nor the doctors taking care of them will be told about the results of the research.

This is an investigational study. CellSearch (the technology used to count circulating tumor cells) is approved by the FDA for breast cancer prognosis. About 660 patients will take part in this multicenter study. About 100 patients will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed invasive breast cancer. Patients must have clinical and/or radiologic evidence of stage IV disease. Tumor may be of any hormone receptor type.
* Patients must have newly diagnosed stage IV breast cancer that is scheduled to start a new systemic therapy.
* Patients may have measurable or non-measurable disease.
* Extent of disease will be determined by physical examination and imaging studies as per the primary physician. The tests utilized may include: (bone scans, PET/CT scans, CT of the abdomen, chest radiograph and/or CT of the chest for visceral metastases, sonogram and/or MRI for soft tissue disease). Patients with skin lesions will have photographs to evaluate their lesions.
* ECOG performance status 0-2.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policies of the hospital. The only acceptable consent form is the one attached at the end of this protocol.

Exclusion Criteria:

* Patients with evidence of local regional recurrence only are excluded.
* Patients who have received prior therapy for their metastatic breast disease.
* Patients with known evidence of brain metastases (unless previously treated or stable) or carcinomatous meningitis.
* Patients with history of any prior malignancies that have not been disease-free for at least 5 years prior to study entry.
* Patients unwilling or unable to give consent.
* Patients unwilling or unable to provided follow-up on their condition.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed stage IV breast cancer scheduled to start systemic therapy.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To detect and count cancer cells in the blood of patients who have recently been diagnosed with a recurrent breast cancer. | 26 Months

SECONDARY OUTCOMES:
To learn if the detection of circulating cancer cells is a predictor for a worse disease prognosis. | 26 Months

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cristofanilli, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org